CLINICAL TRIAL: NCT03745040
Title: Does Liposomal Bupivacaine Improve Postoperative Pain Control After One Level Posterior Spinal Fusion With Instrumentation
Brief Title: Liposomal Bupivacaine in One-level Instrumented Posterior Spinal Fusion
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Allina Health System (Other)
Collaborators: Twin Cities Spine Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1252230
Record Dates: First submitted 2018-11-05; First posted 2018-11-19 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Lumbar Spinal Stenosis; Lumbar Disc Herniation; Lumbar Disc Disease; Lumbar Spondylolisthesis
MeSH Terms: conditions — Spinal Stenosis; Intervertebral Disc Displacement; Intervertebral disc disease; Spondylolisthesis

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized clinical trial with two cohorts: one experimental and one control.
Who Masked: Participant
Masking Description: Subjects will be blinded and will not be informed if they received the study drug or not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Exparel (Experimental): Standard of Care plus Liposomal bupivacaine (Exparel®). Dosage: Exparel® 20 mL single use vial, 1.3% (13.3 mg/mL), Maximum dose of 266 mg (20 mL).
  Frequency: Single intraoperative administration
  Interventions: Drug: Liposomal bupivacaine
- Group B: No Exparel (No Intervention): Standard of Care

INTERVENTIONS:
Drug: Liposomal bupivacaine — 20ml bupivacaine liposome injectable suspension 1.3% (266mg) + 50ml 0.25% Bupivacaine (150mg) + 70ml preservative-free 0.9% neutral saline
  Other Names: Exparel
  Arms: Group A: Exparel

SUMMARY:
This study will describe postoperative pain management for spine surgery patients receiving liposomal bupivacaine (Exparel®) compared to patients not receiving the drug.

DETAILED DESCRIPTION:
This study will describe postoperative pain management for spine surgery patients receiving liposomal bupivacaine (Exparel®) compared to patients not receiving the drug. It is a prospective, randomized clinical trial with two cohorts: Group A: standard of care (SOC) plus liposomal bupivacaine (n=30) and Group B: SOC (n=30). All subjects will undergo open single-level posterior decompression and instrumented fusion for degenerative spondylolisthesis. The surgery is not an experimental procedure. Prior to closing the surgical wound, liposomal bupivacaine will be administered to Group A. The administration of the drug is a study procedure, but note that this is an indicated use of the drug. Postoperatively, subjects will be assessed for pain and opioid consumption. The investigator's hypothesis for statistical analysis is that there will be a 30% decrease in pain medication requirement for the experimental group (Group A: Liposomal bupivacaine ) versus the control group (Group B: No Liposomal bupivacaine).

ELIGIBILITY:
Inclusion Criteria:

* Has a primary diagnosis of single-level lumbar stenosis, disc herniation, and/or spondylolisthesis excluding degenerative disc disease
* Receives open, one-level posterior spinal fusion

Exclusion Criteria:

* Is opioid-tolerant. Opioid tolerant patients are receiving, for one week or longer, at least 60 mg oral morphine/day, 25 mcg transdermal fentanyl/hour, 30 mg oral oxycodone/day, 8 mg oral hydromorphone/day, 25 mg oral oxymorphone/day, or an equianalgesic dose of another opioid.
* Experienced intraoperative complications (i.e., a dural tear or durotomy). Intra- and post-operative data will be excluded from the analysis for these patients.
* Has severe liver disease. Bupivacaine is primarily metabolized in the liver via conjugation with glucuronic acid. Patients with liver disease, especially severe disease may be more susceptible to toxicity.
* Has severe renal disease. Bupivacaine and the metabolite are primarily excreted by the kidneys. Excretion can be significantly changed by urinary perfusion, the presence of renal disease, factors affecting urinary pH, and renal blood flow
* Is less than 18 years old.
* Is pregnant.
* Cannot read and speak English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-26 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Pain Scores | Through study completion, an average of 2.5 days
  Change in Visual Analog Pain Scores over time; respondents report pain at incision site and at drain site on a scale of No pain (0) to Intolerable pain (10).

SECONDARY OUTCOMES:
Number of Participants with Pain | Through study completion, an average of 2.5 days
  Proportion of pain free subjects, an average of 2.5 days
Discomfort | Through study completion, an average of 2.5 days
  Overall Benefit of Analgesia Score. Respondents complete seven questions, each with a score of 0 (minimal or not at all) to 4 (maximum or very much); the total OBAS ranges between 0 (complete relief of pain) and 28 (no benefit).
Total Opioid Consumption | Through study completion, an average of 2.5 days
  Total postsurgical opioid consumption in morphine equivalents
Number of Opioid-related Adverse Events | Through study completion, an average of 2.5 days
  Average number of opioid-related adverse events per patient
Patient Cost of In-Hospital Stay | Through study completion, an average of 2.5 days
  Total combined cost in dollars of hospital room, drugs, laboratory tests, physical therapy, and respiratory therapy
Length of Stay | Through study completion, an average of 2.5 days
  Number of days in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Alcala-Marquez, MD, Principal Investigator — Allina Health System
Locations (2):
- United States (2):
  - Abbott Northwestern Hospital, Allina Health System, Minneapolis, Minnesota
  - United Hospital, Allina Health System, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Vaishya R, Wani AM, Vijay V. Local Infiltration Analgesia reduces pain and hospital stay after primary TKA: randomized controlled double blind trial. Acta Orthop Belg. 2015 Dec;81(4):720-9. PMID 26790796
- [Background] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949
- [Background] Dias AS, Rinaldi T, Barbosa LG. The impact of patients controlled analgesia undergoing orthopedic surgery. Braz J Anesthesiol. 2016 May-Jun;66(3):265-71. doi: 10.1016/j.bjane.2013.06.023. Epub 2015 Apr 17. PMID 27108823
- [Background] McBeath DM, Shah J, Sebastian L, Sledzinski K. The effect of patient controlled analgesia and continuous epidural infusion on length of hospital stay after total knee or total hip replacement. CRNA. 1995 Feb;6(1):31-6. PMID 7599545
- [Background] Chahar P, Cummings KC 3rd. Liposomal bupivacaine: a review of a new bupivacaine formulation. J Pain Res. 2012;5:257-64. doi: 10.2147/JPR.S27894. Epub 2012 Aug 14. PMID 23049275
- [Background] Barrington JW, Olugbode O, Lovald S, Ong K, Watson H, Emerson RH Jr. Liposomal Bupivacaine: A Comparative Study of More Than 1000 Total Joint Arthroplasty Cases. Orthop Clin North Am. 2015 Oct;46(4):469-77. doi: 10.1016/j.ocl.2015.06.003. Epub 2015 Aug 6. PMID 26410636
- [Background] Cherian JJ, Barrington J, Elmallah RK, Chughtai M, Mistry JB, Mont MA. Liposomal Bupivacaine Suspension, Can Reduce Length of Stay and Improve Discharge Status of Patients Undergoing Total Hip Arthroplasty. Surg Technol Int. 2015 Nov;27:235-9. PMID 26680403
- [Background] Chughtai M, Cherian JJ, Mistry JB, Elmallah RD, Bennett A, Mont MA. Liposomal Bupivacaine Suspension Can Reduce Lengths of Stay and Improve Discharge Status of Patients Undergoing Total Knee Arthroplasty. J Knee Surg. 2016 Jul;29(5):e3. doi: 10.1055/s-0036-1584272. Epub 2016 Jun 10. No abstract available. PMID 27285180
- [Background] Emerson RH, Barrington JW, Olugbode O, Lovald S, Watson H, Ong K. Comparison of Local Infiltration Analgesia to Bupivacaine Wound Infiltration as Part of a Multimodal Pain Program in Total Hip Replacement. J Surg Orthop Adv. 2015 Winter;24(4):235-41. PMID 26731387
- [Background] Emerson RH Jr, Barrington JW, Olugbode O, Lovald S, Watson H, Ong K. Femoral Nerve Block Versus Long-Acting Wound Infiltration in Total Knee Arthroplasty. Orthopedics. 2016 May 1;39(3):e449-55. doi: 10.3928/01477447-20160315-03. Epub 2016 Mar 29. PMID 27018607
- [Background] Yu SW, Szulc AL, Walton SL, Davidovitch RI, Bosco JA, Iorio R. Liposomal Bupivacaine as an Adjunct to Postoperative Pain Control in Total Hip Arthroplasty. J Arthroplasty. 2016 Jul;31(7):1510-5. doi: 10.1016/j.arth.2016.01.004. Epub 2016 Jan 21. PMID 26872584
- [Background] Kim KT, Cho DC, Sung JK, Kim YB, Kang H, Song KS, Choi GJ. Intraoperative systemic infusion of lidocaine reduces postoperative pain after lumbar surgery: a double-blinded, randomized, placebo-controlled clinical trial. Spine J. 2014 Aug 1;14(8):1559-66. doi: 10.1016/j.spinee.2013.09.031. Epub 2013 Nov 8. PMID 24216403
- [Background] Puffer RC, Tou K, Winkel RE, Bydon M, Currier B, Freedman BA. Liposomal bupivacaine incisional injection in single-level lumbar spine surgery. Spine J. 2016 Nov;16(11):1305-1308. doi: 10.1016/j.spinee.2016.06.013. Epub 2016 Jun 24. PMID 27349628
- [Background] Tomov M, Tou K, Winkel R, Puffer R, Bydon M, Nassr A, Huddleston P, Yaszemski M, Currier B, Freedman B. Does Subcutaneous Infiltration of Liposomal Bupivacaine Following Single-Level Transforaminal Lumbar Interbody Fusion Surgery Improve Immediate Postoperative Pain Control? Asian Spine J. 2018 Feb;12(1):85-93. doi: 10.4184/asj.2018.12.1.85. Epub 2018 Feb 7. PMID 29503687
- [Background] Wang MY, Grossman J. Endoscopic minimally invasive transforaminal interbody fusion without general anesthesia: initial clinical experience with 1-year follow-up. Neurosurg Focus. 2016 Feb;40(2):E13. doi: 10.3171/2015.11.FOCUS15435. PMID 26828882
- [Background] Kalso E, Edwards JE, Moore AR, McQuay HJ. Opioids in chronic non-cancer pain: systematic review of efficacy and safety. Pain. 2004 Dec;112(3):372-380. doi: 10.1016/j.pain.2004.09.019. PMID 15561393
- [Background] Benyamin R, Trescot AM, Datta S, Buenaventura R, Adlaka R, Sehgal N, Glaser SE, Vallejo R. Opioid complications and side effects. Pain Physician. 2008 Mar;11(2 Suppl):S105-20. PMID 18443635
- [Background] Oderda GM, Evans RS, Lloyd J, Lipman A, Chen C, Ashburn M, Burke J, Samore M. Cost of opioid-related adverse drug events in surgical patients. J Pain Symptom Manage. 2003 Mar;25(3):276-83. doi: 10.1016/s0885-3924(02)00691-7. PMID 12614962
- [Background] Oderda GM, Gan TJ, Johnson BH, Robinson SB. Effect of opioid-related adverse events on outcomes in selected surgical patients. J Pain Palliat Care Pharmacother. 2013 Mar;27(1):62-70. doi: 10.3109/15360288.2012.751956. Epub 2013 Jan 9. PMID 23302094
- [Background] Million R, Hall W, Nilsen KH, Baker RD, Jayson MI. Assessment of the progress of the back-pain patient 1981 Volvo Award in Clinical Science. Spine (Phila Pa 1976). 1982 May-Jun;7(3):204-12. doi: 10.1097/00007632-198205000-00004. PMID 6214028
- [Background] Lehmann N, Joshi GP, Dirkmann D, Weiss M, Gulur P, Peters J, Eikermann M. Development and longitudinal validation of the overall benefit of analgesia score: a simple multi-dimensional quality assessment instrument. Br J Anaesth. 2010 Oct;105(4):511-8. doi: 10.1093/bja/aeq186. Epub 2010 Aug 6. PMID 20693179

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT03745040/Prot_SAP_000.pdf